CLINICAL TRIAL: NCT07028021
Title: Study on Water Turnover of the Chinese Population Based on Deuterium Dilution Method
Status: Recruiting | Type: Observational
Sponsor: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, Xueying Zhang, Principal Investigator, Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Other Study IDs: SIAT-IRB-241115-H0925
Record Dates: First submitted 2025-06-03; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Water Turnover; Population Water Requirements; Deuterium Dilution

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Volunteers from Beijing: A total of 50 local volunteers will be recruited in Beijing to participate in the study. The study procedures will include height measurement, body composition analysis, body water turnover assessment, water intake documentation, physical activity level monitoring, and evaluation of environmental factors (temperature, humidity, and altitude).
- Volunteers from Shenzhen: A total of 50 local volunteers will be recruited in Shenzhen to participate in the study. The study procedures will include height measurement, body composition analysis, body water turnover assessment, water intake documentation, physical activity level monitoring, and evaluation of environmental factors (temperature, humidity, and altitude).
- Volunteers from Shenyang: A total of 50 local volunteers will be recruited in Shenyang to participate in the study. The study procedures will include height measurement, body composition analysis, body water turnover assessment, water intake documentation, physical activity level monitoring, and evaluation of environmental factors (temperature, humidity, and altitude).
- Volunteers from Yantai: A total of 50 local volunteers will be recruited in Yantai to participate in the study. The study procedures will include height measurement, body composition analysis, body water turnover assessment, water intake documentation, physical activity level monitoring, and evaluation of environmental factors (temperature, humidity, and altitude).
- Volunteers from Xining: A total of 50 local volunteers will be recruited in Xining to participate in the study. The study procedures will include height measurement, body composition analysis, body water turnover assessment, water intake documentation, physical activity level monitoring, and evaluation of environmental factors (temperature, humidity, and altitude).
- Volunteers from Wenzhou: A total of 50 local volunteers will be recruited in Wenzhou to participate in the study. The study procedures will include height measurement, body composition analysis, body water turnover assessment, water intake documentation, physical activity level monitoring, and evaluation of environmental factors (temperature, humidity, and altitude).

SUMMARY:
Water is essential for sustaining life and maintaining health. The human body relies on water to transport nutrients and waste products, lubricate joints, regulate body temperature, and preserve tissue structure. International research has shown that losing just 2% of body weight through water loss can impair physiological functions and reduce response capacity. Adequate water intake plays a crucial protective role in health: it helps regulate body weight, lowers the risk of chronic diseases such as cardiovascular and cerebrovascular conditions, and supports cognitive function.

However, the common recommendation to drink eight cups of water per day lacks strong scientific evidence. Most national hydration guidelines are based on average population intake, and personalized water intake recommendations have yet to be fully developed.

In this study, the investigators will use the deuterium dilution technique to measure water turnover in volunteers. Body composition will be assessed using the TANITA MC-780, while a seven-day fluid intake diary will track daily water consumption. Physical activity levels will be monitored using GT3 devices, and environmental data-including altitude, temperature, and humidity-will be collected based on participants' locations.

The goal of this study is to collect comprehensive data on the physiological traits, environmental influences, and hydration needs of the Chinese population. This will allow for refinement and optimization of current prediction equations for water requirements. Ultimately, the investigators aim to develop a new, individualized water intake algorithm tailored to the Chinese population by quantifying the proportion of water intake relative to total water requirements.

DETAILED DESCRIPTION:
The following assessments will be conducted with the volunteers:

Height Measurement: Height will be measured using a Seca 217 stable stadiometer. Participants will be asked to remove their shoes for the measurement.

Body Composition Measurement: Body composition will be assessed using the TANITA MC-780 device. This provides individual segmental weight measurements for the right arm, left arm, trunk, right leg, and left leg. A comprehensive report will also be generated, including body weight (BW), body fat percentage (fat%), fat mass (FM), body mass index (BMI), and fat-free mass (FFM).

Body Water Measurement: Total body water will be measured using the deuterium dilution technique. Participants will arrive at the laboratory after an overnight fast and provide a baseline urine sample. They will then ingest a dose of deuterated water calculated based on their body weight. Additional urine samples will be collected three and four hours after dosing. The increase in deuterium concentration compared to baseline will be used to calculate total body water.

Physical Activity Measurement: Physical activity will be monitored using a GT3 accelerometer, worn near the hip for seven consecutive days. The device should be removed during bathing or swimming. The first day of data will be excluded, as well as any day with less than 12 hours of wear time. Valid data must include at least two weekdays and two weekend days.

Water Intake Measurement: Water intake will be tracked using a seven-day liquid intake diary. Participants will be provided with a form to record the type, time, and amount of liquid consumed across eight specific time intervals each day. Detailed instructions will be provided. Continuous recording for the full seven-day period is required.

Environmental Data Collection: Environmental temperature and relative humidity will be recorded using an iButton device. The average altitude of each participant's city of residence will be determined using GPS-based altitude software.

ELIGIBILITY:
Inclusion Criteria:

1. Stable body weight over the past year
2. Ability to perform normal physical activities

Exclusion Criteria:

1. History of chronic diseases such as diabetes, liver disease, kidney disease, or any other conditions that may affect fluid metabolism
2. Use of diuretics or other medications that influence urine output
3. Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of healthy individuals with stable body weight over the past year and the ability to engage in normal physical activities. Participants had no history of chronic diseases, were not taking diuretics or other medications that affect urine output, and female participants were neither pregnant nor breastfeeding.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Height | Height measurement will be conducted on the first day of the study for each volunteer and will take approximately 2 minutes.
  Height in meters (m) will be measured using the SECA 217 stable stadiometer. Subjects will be measured without shoes.
Body weight | Body weight will be conducted on the first day of the study for each volunteer and will take approximately 5 minutes.
  Body weight in kilograms (kg) will be measured using the TANITA MC-780 device. Participants will be barefoot and dressed in light clothing during the measurement.
Body composition | Body composition ( fat mass )will be conducted on the first day of the study for each volunteer and will take approximately 5 minutes.
  The TANITA (TANITA MC-780) device will be used to measure fat mass (in kilograms, kg) as a primary indicator of body composition. Participants will be asked to remove all metal accessories and wear light clothing during the measurement.
Body water | Deuterium dilution technology will be initiated at the start of the volunteer's research visit, with each volunteer undergoing a one-week data collection period .
  Body water in kilograms will be measured by deuterium dilution. Subjects will attend the lab after an overnight fast and provide a baseline urine sample. They will then drink a dose of deuterated water based on their body weight. Urine samples will be collected at 4 hours after dosing, and 7 days after dosing, to measure the level of deuterium isotope in the body relative to the baseline. The increase in deuterium concentration allows for the calculation of total body water based on the dilution principle.
Physical Activity | Physical activity will be initiated at the start of the volunteer's research visit, with each volunteer undergoing a one-week data collection period.，and will be used in subsequent data analyses.
  Physical activity (in vector magnitude counts) of the participants will be recorded using GT3X accelerometer worn near the hip for a consecutive period of 7 days. The monitor should not be worn while bathing or swimming. The first day is discarded along with any day where the wear time is less than 12 hours. For a valid measure the goal is to get 2 weekday and 2 weekend days.
Water Intake Measurement | Water intake will be initiated at the start of the volunteer's research visit, with each volunteer undergoing a one-week data collection period, and will be used in subsequent data analyses.
  Water intake will be recorded using a seven-day liquid intake diary. A standardized form will be provided to the volunteers, where they will record the type, time, and amount (in milliliters, mL) of liquid consumed across approximately four specific time periods each day. Detailed recording standards and instructions will be included in the form.
Environmental temperature | Environmental temperature exposure will be monitored for one week beginning at the start of the volunteer's research visit
  The iButton (DS1921G) will be used to assess the subject's exposure to temperature (in Degrees Celsius) by measuring both indoor and outdoor temperatures. The devices will be placed on the subject's hand bag or clothes, the indoor wall of the home and workplace, and the exterior building surface.
Average residential altitude of participant | The average altitude will be recorded at the start of the volunteer's participation in the study and will take approximately 2 minutes.
  The average altitude (in meters) of the participant's residential city will be determined using GPS-based altitude software.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing, Beijing, Beijing Municipality, China